CLINICAL TRIAL: NCT00334022
Title: A Pilot Randomized Controlled Trial of Adding Enfuvirtide to Standard Combination Antiretroviral Therapy in HIV-infected Individuals With Full Virologic Suppression to Further Suppress Proviral HIV DNA
Brief Title: Fuzeon Viral Decay Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Immunodeficiency Research Collaborative (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Roche-FVD-1
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: HIV-1
Keywords: Fuzeon; Viral Decay
MeSH Terms: interventions — Enfuvirtide

ARMS (2):
- Did not receive enfuvirtide (Placebo Comparator): patients were randomized to either receive enfuviratide or not receive it
  Interventions: Drug: enfuvirtide
- enfuvirtide (Active Comparator): enfuvirtide 1ml BID
  Interventions: Drug: enfuvirtide

INTERVENTIONS:
Drug: enfuvirtide — 1ml BID

SUMMARY:
In order to better understand the source(s) and the mechanism(s) of HIV persistence and to potentially lead to further suppression of HIV from viral reservoirs, we propose to examine the effect of co-administration of enfuvirtide, an entry inhibitor of HIV, on diminution of the size of the viral reservoir in infected individuals who are receiving effective antiviral therapy for extended periods of time (> 5 years).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be HIV infected
2. Patient must be > 18 years old
3. Patient must be taking standard combination antiretroviral therapy with 2-3 NRTIs and 1-2 PIs or a NNRTIs for at least five years
4. Patient must have a viral load < 50 copies/mL (using the standard available methods of detection) during the entire time on standard combination antiretroviral therapy except for initial fall of viral load
5. Patient must have a CD4 count above 400 cells/mm3 in last 3 months
6. Female patient must agree to use two methods of birth control or abstinence during the period of the study
7. Patient has to have signed full informed consent

Exclusion Criteria:

1. Patient who would have difficulty participating in a trial due to non-adherence or substance abuse
2. Patient who have taken mono or dual antiretroviral therapy
3. Patient who have had a viral load > 50 copies/mL on any antiretroviral regimen
4. Patient with any of the following abnormal laboratory test results in screening:

   * Hemaglobin < 100 g/L
   * Neutrophil count < 750 cells/uL
   * Platelet count < 50,000 cells/L
   * AST or ALT > 5X the upper limit of normal
   * Creatinine > 250 umol/L
5. Patient with a malignancy
6. Patient with other significant underlying disease (non-HIV) that might impinge upon disease progression or death
7. Patient with an active AIDS-defining illnesses in the past six months
8. Patients who are pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The change of proviral HIV-1 DNA in both purified resting and activated CD4 T cells from baseline to month 6. | 6 months
  The change of proviral HIV-1 DNA in both purified resting and activated CD4 T cells from baseline to month 6.

SECONDARY OUTCOMES:
To determine the change of proviral HIV-1 DNA from baseline to month 3 | 3 months
  To determine the change of proviral HIV-1 DNA from baseline to month 3
To determine the change of proviral HIV-1 DNA from months 6 to 9 after the enfurvitide has been stopped for 3 months in the treatment arm | 9 months
  To determine the change of proviral HIV-1 DNA from months 6 to 9 after the enfurvitide has been stopped for 3 months in the treatment arm
To quantify plasma HIV (limit of detection 2 copies/ml of plasma) | 9 months
  To quantify plasma HIV (limit of detection 2 copies/ml of plasma)
To quantify cell associated HIV RNA (unspliced and multiply spliced) in resting and activated CD4+ T cells | 9 months
  To quantify cell associated HIV RNA (unspliced and multiply spliced) in resting and activated CD4+ T cells
To determine the decay characteristics of HIV in resting CD4+ T cells by quantitative co-culture assays | 9 months
  To determine the decay characteristics of HIV in resting CD4+ T cells by quantitative co-culture assays
To determine the half-life of HIV in resting CD4+ T cells | 9months
  To determine the half-life of HIV in resting CD4+ T cells
To carry out phylogenetic analysis of HIV in the plasma, resting, and activated CD4+ T cell compartments | 9 months
  To carry out phylogenetic analysis of HIV in the plasma, resting, and activated CD4+ T cell
To quantify the amount of HIV in gastrointestinal-associated lymphoid tissue (GALT) by quantitative co-culture assays (as part of a sub-study - see GALT sub-study) | 9 months
  To quantify the amount of HIV in gastrointestinal-associated lymphoid tissue (GALT) by quantitative co-culture assays (as part of a sub-study - see GALT sub-study)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Kovacs, MD, Principal Investigator — University of Toronto
Locations (1):
- Maple Leaf Medical Clinic, Toronto, Ontario, Canada